CLINICAL TRIAL: NCT07038148
Title: Exploring the Efficacy of Single-stage Stapled Conversion of Gastric Bypass to Sleeve Gastrectomy, More Leak?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Abdelsalam M, Associate Professor of General and Laparoscopic Surgery, Kasr El Aini Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N-8-2025
Record Dates: First submitted 2025-01-25; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-01

CONDITIONS: the Focus of the Study is to Assees Efficacy of Stapled Revision of Gastric Bypass to Sleeve Gastrectomy

STUDY DESIGN:
Intervention Model Description: This is a prospective single-arm clinical trial that will include patients who had gastric bypass done - both RYGB and OAGB-, who developed complications of bypass and are candidates for reversal, but still keen to keep weight loss or even add more weight loss.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Candidates of several of bypass to sleeve (Experimental): This interventional study with a single arm assesses the effectiveness and safety of converting gastric bypass to sleeve gastrectomy using a laparoscopic stapling technique in adults who have complications from earlier gastric bypass procedures. The approach entails closing the prior gastrojejunostomy and performing a sleeve gastrectomy with a stapling method. The outcomes measured will include enhancements in nutritional status, weight regain, quality of life, and symptoms of GERD over a follow-up period of 6 months.
  Interventions: Procedure: Stapled reversal of gastric bypass to sleeve gastrectomy utilising stapling technique.

INTERVENTIONS:
Procedure: Stapled reversal of gastric bypass to sleeve gastrectomy utilising stapling technique. — This research entails a single-stage laparoscopic conversion of gastric bypass to sleeve gastrectomy. The procedure entails the closure of the gastrojejunostomy with an endo-stapler and the reconstruction of the stomach by resecting along the greater curvature to create a sleeve gastrectomy. An intraoperative leak test will be conducted using methylene blue. Patients are monitored postoperatively for at least 24 hours, with subsequent assessments of nutritional status, weight, gastroesophageal reflux disease (GERD) symptoms, and quality of life at 3 and 6 months.

SUMMARY:
Laparoscopic gastric bypass - including both Roux-en-Y gastric bypass (RYGB) and one anastomosis gastric bypass (OAGB) - is one of the most frequently performed procedures. However, as the number of gastric bypass surgeries increases, complications are being reported more often. While most post-bypass complications can be managed non-surgically, a small number of persistent cases may require a reversal to normal anatomy or conversion to another procedure.

Many patients who experience severe complications from gastric bypass are reluctant to undergo a reversal to normal anatomy due to fears of regaining weight. As a result, converting to another type of surgery becomes a more logical alternative.

Complications requiring conversion are numerous and negatively affect the quality of life, such as retrograde intussusception, weight regain, intractable dumping syndrome, and nutritional deficiencies. The high cost of obligatory postoperative vitamins is a potential cause of conversion especially in low-income countries.

The conversion procedure is technically demanding and has a relatively higher rate of postoperative complications, making it less commonly performed. Additionally, limited data is available regarding the procedure and its long-term outcomes, making it an unexplored sea of hope for people who wish to manage intractable complications of gastric bypass and maintain weight loss.

DETAILED DESCRIPTION:
Objectives: To study efficacy, safety, and patient outcomes following laparoscopic gastric bypass conversion to sleeve gastrectomy.

Study population & Sample size :

Adult patients undergoing single-stage laparoscopic stapled conversion of gastric bypass to sleeve gastrectomy in Kasr Alainy Sample size: 11 patients Study Design: This is a prospective single-arm clinical trial.

Methods: Patients who will attend our bariatric outpatient clinic will be enlisted according to inclusion criteria. A detailed history of anthropometric measures, chronic diseases, and previous surgeries will be recorded. After patient education, preoperative routine labs and imaging will be performed.

A preoperative 3D gastric volumetry CT scan will be performed to all patients included in this study.

The procedure will consist of converting the gastric bypass to a sleeve gastrectomy using a stapling technique.

The average length of hospital stay will be included. Follow up of nutritional status will be done using laboratory parameters (Hb, Ferritin, Vitamin D, Zn, Mg, serum Albumin, Calcium) in 3 months and 6 months postoperatively, quality of life will be assessed using bariatric quality of life index in 3 months and 6 months postoperatively.

Patient weight will be documented monthly to evaluate weight regain, GERD symptoms will be assessed using GERD score in 3 months and 6 months postoperatively.

Possible Risk (s) to study population:

1. Postoperative pain.
2. Postoperative nausea and vomiting.
3. Bleeding
4. Anastomotic leakage
5. Stricture

Outcome parameters:

* Primary outcomes

  1. Improvement of nutritional status.
  2. Weight regain.
* Secondary outcome parameters

  1. Quality of life
  2. GERD symptoms

Statistical analysis plan:

Data analysis packages will be SPSS version 21. Qualitative data will be presented by number and percentage, quantitative data will be presented by mean, standard deviation, median, and interquartile range.

Parametric and non-parametric tests of significant will be done (chi-square, student t-test, and Mann-Whitney test).

Correlation analysis tests and regression will be done. The level of significance was set at p equal to or below 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-70
* Adult patients undergoing single-stage laparoscopic stapled conversion of gastric bypass to sleeve gastrectomy.
* Patients accept to sign an informed consent and will commit to follow-up.

Exclusion Criteria:

* Patients with reversal gastric bypass to normal anatomy.
* Patient with uncontrolled systemic disease.
* Patients with active psychological disorders.
* Patients with active substance abuse.
* Patients with intra-operative technical difficulties hindering the conversion of gastric bypass to sleeve gastrectomy.
* Patients refusing to sign an informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Nutritional Status | one year
  nutritional status of patient will be assessed by general examination, assessment of lower limb edema, serum albumin and hemoglobin
Weight Regain | one year
  The initial weight at the time of the procedure will be measured in kg, and at follow-up, it will be reassessed at three, six, and twelve months. Weight assessment will be part of the BMI assessment in kg/m2

SECONDARY OUTCOMES:
Quality of Life | one year
  The Short Form 36 (SF-36) questionnaire will be used to assess quality of life and overall health status.
GERG symptoms | One year
  GERD symptoms will be assessed at three, six, and twelve months of follow-up. The GERD-Health Related Quality of Life (GERD-HRQL) Questionnaire will be used in this study.

OTHER OUTCOMES:
Possible Risks | One year
  1. Post operative pain.
  2. Post operative nausea and vomiting.
  3. Bleeding
  4. Anastomotic leakage
  5. Stricture

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy Medical School, Cairo University, Cairo, Old Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Okut G, Turgut E, Kaplan K, Sumer F, Kayaalp C. Can revision of RYGB to sleeve gastrectomy be a solution to inadequate weight loss treatment? Cir Cir. 2022;90(S1):25-30. doi: 10.24875/CIRU.21000458. PMID 35944120
- [Background] Sjostrom L, Lindroos AK, Peltonen M, Torgerson J, Bouchard C, Carlsson B, Dahlgren S, Larsson B, Narbro K, Sjostrom CD, Sullivan M, Wedel H; Swedish Obese Subjects Study Scientific Group. Lifestyle, diabetes, and cardiovascular risk factors 10 years after bariatric surgery. N Engl J Med. 2004 Dec 23;351(26):2683-93. doi: 10.1056/NEJMoa035622. PMID 15616203